CLINICAL TRIAL: NCT05814991
Title: A Cohort Prospective Study of Predictors Influencing the Quality of Visualization of the Operating Field During Orthognathic Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia (Other)
Responsible Party: Sponsor
Other Study IDs: NMSC-01-23
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Malocclusion; Maxillofacial Injuries; Orthodontics; Hemorrhage
Keywords: nitroglycerin; the quality of visualization of the operating field; Near-infrared Spectroscopy (NIRS); cerebral oximetry; regional cerebral oxygen saturation (rSO2); Le Fort; I; controlled hypotension anesthesia
MeSH Terms: conditions — Malocclusion; Maxillofacial Injuries; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing bimaxillary osteotomy under general anesthesia
  Interventions: Drug: Nitroglycerin solution; Device: monitoring of cerebral oxygen saturation

INTERVENTIONS:
Drug: Nitroglycerin solution — Controlled hypotension will be induced (intravenous administration of nitroglycerin 2-10 µg/kg/min) 15 minutes prior to the start of mucosal detachment, and will be sustained for the osteotomy stage.
Device: monitoring of cerebral oxygen saturation — NIRS-based monitoring of rSO2 has unique advantages: directly or indirectly detecting physiological changes and metabolic processes, it is easy to realize, and involves simple procedures.
  Other Names: NIRS

SUMMARY:
It is very important to decrease the bleeding during bimaxillary osteotomy in order to increase the visibility of the surgical site. Our primary goal is to investigate the predictive value of pre- and perioperative factors, including controlled hypotension, on visibility of surgical site during bimaxillary osteotomy.

DETAILED DESCRIPTION:
100 patients undergoing bimaxillary osteotomy under general anesthesia will be included into this prospective cohort study.

There will be two episodes of controlled hypotension for upper and lower jaw respectively. Hypotension will be induced and sustained according to the same procedure as described here. Controlled hypotension will be induced (intravenous administration of nitroglycerin 2-10 µg/kg/min) 15 minutes prior to the start of mucosal detachment, and will be sustained for the osteotomy stage. The surgeon will evaluate the surgical field quality (in terms of bleeding) according to Modena Bleeding Score (MBS), with scores 1-2 being satisfactory to proceed with the osteotomy. The following arterial pressure correction (proceeding with controlled hypotension or returning to normotension) will depend on the bleeding in the surgical field and the monitoring of cerebral oxygen saturation carried out using near-infrared spectroscopy (NIRS) . The lowest targeted arterial pressure in order to have a clear surgical field will be 55 mmHg. However when the cerebral oxygen saturation decreases by 20% compared with the baseline at any arterial pressure level intervention would be carried out by Norepinephrine (intravenous, individual dosage for each patient - as judged by the anesthesiologist). Arterial blood samples will be taken at 3 time points (at the start of the surgery, during controlled hypotension phase, after extubation) for arterial gas analysis. Two blood samples will be taken to measure (prior to surgery and immediately after surgery) neuron-specific enolase (NSE), cystatin c and troponin I levels. The general condition, operation, anesthesia and hospitalization related data of the patients will be recorded. Cognitive function will be evaluated within 3 days before surgery and 2 days and 1 month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients refered for bimaxillary osteotomy under general anesthesia with endotracheal intubation;
* Anesthesia risk classes (ASA) I and II;
* Written statement of informed consent.

Exclusion Criteria:

* Hypertension as a symptom of hypertensive heart disease or endocrine dysfunction;
* Patients receiving antihypertensive drugs;
* Patients receiving anticoagulant therapy;
* Ischemic heart disease;
* Cerebrovascular insufficiency;
* Severe hypovolemia;
* Anemia;
* BMI 30 kg/m2 and higher;
* Connective tissue disorders;
* Pregnancy;
* Participation in other clinical studies;
* Recent history of substance abuse (recreational drugs, alcohol);
* Allergies to drugs used in the study;
* Anxiety requiring psychiatrist supervision and pharmacological therapy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients undergoing bimaxillary osteotomy under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Visibility of surgical site | during osteotomy, up to 90 minutes
  Surgical site will be rated according to Modena Bleeding Score (MBS) by the same surgeon in terms of bleeding during osteotomy. The MBS goes from Grade 1 - no bleeding to Grade 5 - bleeding that prevents every surgical procedure except those dedicated to bleeding control.

SECONDARY OUTCOMES:
Proportion of patients with cerebral desaturation | during osteotomy, up to 90 minutes
  Proportion of patients with decrease in cerebral oxygen saturation decreased by 20% compared with the baseline for 300 seconds without improvement
changes in the values of mean arterial pressure | during the whole surgery (from start to finish - the timing stated in the surgery protocol)
  Changes in mean arterial pressure (MAP) values before and during controlled hypotension phase will be registered.
  MAP calculated as follows:
  MАP = Diastolic blood pressure + ((Systolic blood pressure - Diastolic blood pressure) / 3).
Changes in neuron-specific enolase (NSE) concentration | 3 time-points during the surgery - immediately after anesthesia induction, at the time of controlled hypotension (5 minutes after induction of controlled hypotension, i.e. nitroglycerin i.v. administration), immediately after extubation
  NSE is released from neurons during injury and it's high blood concentration is associated with ischemic brain injury. Level of NSE will be measured in blood samples taken during surgery. Increase of NSE level suggests brain ischemia.
Intraoperative blood loss | during the whole surgery (from start to finish - the timing stated in the surgery protocol)
  Total volume of blood loss during the time of surgery, calculated using direct volumetric measurement.
Cognitive status change | within 3 days before operation, 2 days after surgery, 1 month after surgery
  Cognitive function will be evaluated by means of Mini Mental State Examination (MMSE), which is a 30-point test, validated and commonly used to measure cognitive impairment. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.
Changes in cystatin C concentration | at the start of the surgery, during controlled hypotension phase, immediately after extubation
  Cystatin C is a well investigated biomarker with clear advantages over serum creatinine in patients with extremes in muscle mass, weight, age, and other areas where estimating equations using creatinine have well documented limitations. Increase of cystatin C level suggests kidney impairment.
Change in Troponin I concentration | at the start of the surgery, during controlled hypotension phase, immediately after extubation
  The test can be used to aid in diagnosing myocardial infarction.

CONTACTS AND LOCATIONS:
Locations (1):
- Pirogov National Medical and Surgical Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 6 months after completion of the study
Access Criteria: upon the request

REFERENCES:
- [Background] Pineiro-Aguilar A, Somoza-Martin M, Gandara-Rey JM, Garcia-Garcia A. Blood loss in orthognathic surgery: a systematic review. J Oral Maxillofac Surg. 2011 Mar;69(3):885-92. doi: 10.1016/j.joms.2010.07.019. Epub 2010 Dec 31. PMID 21195531
- [Background] Sugahara K, Koyama Y, Koyachi M, Watanabe A, Kasahara K, Takano M, Katakura A. A clinico-statistical study of factors associated with intraoperative bleeding in orthognathic surgery. Maxillofac Plast Reconstr Surg. 2022 Feb 25;44(1):7. doi: 10.1186/s40902-022-00336-8. PMID 35212834
- [Background] Salma RG, Al-Shammari FM, Al-Garni BA, Al-Qarzaee MA. Operative time, blood loss, hemoglobin drop, blood transfusion, and hospital stay in orthognathic surgery. Oral Maxillofac Surg. 2017 Jun;21(2):259-266. doi: 10.1007/s10006-017-0626-1. Epub 2017 May 2. PMID 28466191
- [Background] Ha TN, van Renen RG, Ludbrook GL, Valentine R, Ou J, Wormald PJ. The relationship between hypotension, cerebral flow, and the surgical field during endoscopic sinus surgery. Laryngoscope. 2014 Oct;124(10):2224-30. doi: 10.1002/lary.24664. Epub 2014 Apr 22. PMID 24604576
- [Background] Ferri J, Druelle C, Schlund M, Bricout N, Nicot R. Complications in orthognathic surgery: A retrospective study of 5025 cases. Int Orthod. 2019 Dec;17(4):789-798. doi: 10.1016/j.ortho.2019.08.016. Epub 2019 Sep 5. PMID 31495753
- [Background] Degoute CS. Controlled hypotension: a guide to drug choice. Drugs. 2007;67(7):1053-76. doi: 10.2165/00003495-200767070-00007. PMID 17488147
- [Background] Ettinger KS, Yildirim Y, Weingarten TN, Van Ess JM, Viozzi CF, Arce K. Hypotensive Anesthesia Is Associated With Shortened Length of Hospital Stay Following Orthognathic Surgery. J Oral Maxillofac Surg. 2016 Jan;74(1):130-8. doi: 10.1016/j.joms.2015.05.025. Epub 2015 May 28. PMID 26047710
- [Background] Lin S, McKenna SJ, Yao CF, Chen YR, Chen C. Effects of Hypotensive Anesthesia on Reducing Intraoperative Blood Loss, Duration of Operation, and Quality of Surgical Field During Orthognathic Surgery: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Oral Maxillofac Surg. 2017 Jan;75(1):73-86. doi: 10.1016/j.joms.2016.07.012. Epub 2016 Jul 25. PMID 27542543
- [Background] Varol A, Basa S, Ozturk S. The role of controlled hypotension upon transfusion requirement during maxillary downfracture in double-jaw surgery. J Craniomaxillofac Surg. 2010 Jul;38(5):345-9. doi: 10.1016/j.jcms.2009.10.012. Epub 2009 Nov 12. PMID 19913434
- [Background] Rodrigo C. Induced hypotension during anesthesia with special reference to orthognathic surgery. Anesth Prog. 1995;42(2):41-58. PMID 8934953
- [Background] Wesselink EM, Kappen TH, Torn HM, Slooter AJC, van Klei WA. Intraoperative hypotension and the risk of postoperative adverse outcomes: a systematic review. Br J Anaesth. 2018 Oct;121(4):706-721. doi: 10.1016/j.bja.2018.04.036. Epub 2018 Jun 20. PMID 30236233
- [Background] Mathis MR, Naik BI, Freundlich RE, Shanks AM, Heung M, Kim M, Burns ML, Colquhoun DA, Rangrass G, Janda A, Engoren MC, Saager L, Tremper KK, Kheterpal S, Aziz MF, Coffman T, Durieux ME, Levy WJ, Schonberger RB, Soto R, Wilczak J, Berman MF, Berris J, Biggs DA, Coles P, Craft RM, Cummings KC, Ellis TA 2nd, Fleishut PM, Helsten DL, Jameson LC, van Klei WA, Kooij F, LaGorio J, Lins S, Miller SA, Molina S, Nair B, Paganelli WC, Peterson W, Tom S, Wanderer JP, Wedeven C; Multicenter Perioperative Outcomes Group Investigators. Preoperative Risk and the Association between Hypotension and Postoperative Acute Kidney Injury. Anesthesiology. 2020 Mar;132(3):461-475. doi: 10.1097/ALN.0000000000003063. PMID 31794513
- [Background] Gregory A, Stapelfeldt WH, Khanna AK, Smischney NJ, Boero IJ, Chen Q, Stevens M, Shaw AD. Intraoperative Hypotension Is Associated With Adverse Clinical Outcomes After Noncardiac Surgery. Anesth Analg. 2021 Jun 1;132(6):1654-1665. doi: 10.1213/ANE.0000000000005250. PMID 33177322
- [Background] Farah GJ, de Moraes M, Filho LI, Pavan AJ, Camarini ET, Previdelli IT, Coelho L. Induced hypotension in orthognathic surgery: a comparative study of 2 pharmacological protocols. J Oral Maxillofac Surg. 2008 Nov;66(11):2261-9. doi: 10.1016/j.joms.2008.06.045. PMID 18940490
- [Background] Rhee SH, An JS, Seo KS, Karm MH. Predictors of Red Blood Cell Transfusion in Bimaxillary Orthognathic Surgery: A Retrospective Study. Int J Med Sci. 2021 Jan 29;18(6):1432-1441. doi: 10.7150/ijms.55567. eCollection 2021. PMID 33628100
- [Background] Thiele RH, Shaw AD, Bartels K, Brown CH 4th, Grocott H, Heringlake M, Gan TJ, Miller TE, McEvoy MD; Perioperative Quality Initiative (POQI) 6 Workgroup. American Society for Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement on the Role of Neuromonitoring in Perioperative Outcomes: Cerebral Near-Infrared Spectroscopy. Anesth Analg. 2020 Nov;131(5):1444-1455. doi: 10.1213/ANE.0000000000005081. PMID 33079868